CLINICAL TRIAL: NCT06821113
Title: Vale+ Tu Salud: Corner-Based Randomized Trial to Test a Latino Day Laborer Program Adapted to Prevent COVID 19
Brief Title: Vale+Tú Salud: Corner-Based Trial to Test a Latino Day Laborer Program Adapted to Prevent COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Maria Eugenia Fernandez-Esquer, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-20-1389 (Phase 3); 1R01MD016328-01 (NIH)
Record Dates: First submitted 2025-02-07; First posted 2025-02-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: Latino Day Laborers
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Cluster Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Group Problem Solving and booster call (Experimental)
  Interventions: Behavioral: COVID-19 Group Problem Solving; Behavioral: Standard of Care; Behavioral: Booster session
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: COVID-19 Group Problem Solving — Participants will have three core components to be delivered at the corner by trained data collectors. Interactive dialogue component that incorporates popular education activities aimed at developing social cohesion among LDLs, building awareness about COVID-19 risks and protective behaviors and developing a personal commitment called "Mi Promesa" to implement COVID mitigation practices. Navigation Component will consist of providing information and linking LDLs with social service providers and the "Multiplicador de salud"/Health Multiplier component that builds from the theoretical and practice-based method of mobilizing social networks and social support.
  Arms: COVID-19 Group Problem Solving and booster call
Behavioral: Standard of Care — Participants will receive a COVID-19 prevention flyer and social resources list only
Behavioral: Booster session — Participants in this group will also receive a "booster phone call" 10 to 15 days after the small group intervention to provide brief prompts to encourage participants to act on their personal commitments and encourage them to seek community resources.
  Arms: COVID-19 Group Problem Solving and booster call

SUMMARY:
The purpose of this study is to determine the cultural, socioeconomic, inter/personal and work-related factors that influence COVID 19 mitigation practices including social distancing, hand-washing and Personal protective equipment (PPE) use, to adapt, implement, and test Vale+Tú Salud in a cluster randomized trial to assess the extent to which LDL report increased adherence with COVID 19 mitigation practices 1 month post intervention and to promote Vale+Tú Salud just-in-time results and increase its capacity to rapidly disseminate findings among groups that serve LDL and other Latino immigrants.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic or Latino
* Be present at the corner for the purposes of looking for work

Exclusion Criteria:

* Have not been previously hired to work at a corner
* Symptoms of COVID-19 in the previous 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in COVID-19 vaccination status as assessed by a survey | Baseline, 4 weeks post intervention
Change in hand washing frequency as assessed by a survey | Baseline, 4 weeks post intervention
Percentage of participants who report contacting the gold card agency | Baseline, 4 weeks post intervention
Percentage of participants who report contacting the agency for assistance to get food | Baseline, 4 weeks post intervention
Percentage of participants who report contacting the agency for assistance for health care resources | Baseline, 4 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Fernandez-Esquer, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No